CLINICAL TRIAL: NCT00330785
Title: An International, Multicentre, Open Label Study To Assess The Effectiveness Of Amlodipine -Atorvastatin Combination In Subjects With Hypertension and Dyslipidaemia. (The JEWEL Study)
Brief Title: Open Label Study Assessing Effectiveness Of Amlodipine/Atorvastatin In Subjects With Hypertension and Dyslipidaemia
Acronym: JEWEL I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3841018
Record Dates: First submitted 2006-02-28; First posted 2006-05-29 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Hypertension; Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — amlodipine, atorvastatin drug combination

INTERVENTIONS:
Drug: Amlodipine/Atorvastatin

SUMMARY:
To evaluate the effectiveness of amlodipine/atorvastatin therapy by assessing the percentage of subjects who reach target blood pressure (BP) and LDL-C targets as defined by their governing guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are above target LDL-C and BP who are eligible for treatment

Exclusion Criteria:

* High liver enzymes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250
Dates: Start 2004-10; Study Completion 2005-09

PRIMARY OUTCOMES:
To evaluate the number of patients who reach target blood pressure (BP) and
LDL-C targets as defined by their governing guidelines.

SECONDARY OUTCOMES:
To assess changes from baseline to end of treatment for the following efficacy
parameters: LDL-C, total cholesterol (TC), triglycerides, high-density lipoprotein
cholesterol (HDL-C), HDL-C/LDL-C ratio, TC/HDL-C ratio. Systolic Blood Pressure
(SBP) and Diastolic Blood Pressue (DBP).

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (95):
- Canada (47):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Red Deer, Alberta
  - Pfizer Investigational Site, Campbell River, British Columbia
  - Pfizer Investigational Site, Chilliwack, British Columbia
  - Pfizer Investigational Site, New Westminster, British Columbia
  - Pfizer Investigational Site, North Vancouver, British Columbia
  - Pfizer Investigational Site, Quesnel, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Antigonish, Nova Scotia
  - Pfizer Investigational Site, Digby, Nova Scotia
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Truro, Nova Scotia
  - Pfizer Investigational Site, Wolfville, Nova Scotia
  - Pfizer Investigational Site, Alymer, Ontario
  - Pfizer Investigational Site, Corunna, Ontario
  - Pfizer Investigational Site, Exeter, Ontario
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Kingston, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, North York, Ontario
  - Pfizer Investigational Site, Oshawa, Ontario
  - Pfizer Investigational Site, Peterborough, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Waterloo, Ontario
  - Pfizer Investigational Site, Weston, Ontario
  - Pfizer Investigational Site, Whitby, Ontario
  - Pfizer Investigational Site, Charlottetown, Prince Edward Island
  - Pfizer Investigational Site, Bonaventure, Quebec
  - Pfizer Investigational Site, Chomedy, Quebec
  - Pfizer Investigational Site, Gatineau, Quebec
  - Pfizer Investigational Site, Granby, Quebec
  - Pfizer Investigational Site, Longueuil, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Saint-Jérôme, Quebec
  - Pfizer Investigational Site, Saint-Lambert, Quebec
  - Pfizer Investigational Site, Saint-Marc-des-Carrieres, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, St-Georges Ouest, Quebec
  - Pfizer Investigational Site, Ste-foy, Quebec
  - Pfizer Investigational Site, Regina, Saskatchewan
  - Pfizer Investigational Site, Rimouski
  - Pfizer Investigational Site, St-Gedeon Beauce
  - Pfizer Investigational Site, St. John's
- United Kingdom (47):
  - Pfizer Investigational Site, Ayr, Ayrshire
  - Pfizer Investigational Site, Sandy, Bedfordshire
  - Pfizer Investigational Site, Peterborough, Cambs
  - Pfizer Investigational Site, Thornhill, Cardiff
  - Pfizer Investigational Site, Fowey, Cornwall
  - Pfizer Investigational Site, Darlington, County Durham
  - Pfizer Investigational Site, Paignton, Devon
  - Pfizer Investigational Site, Plymouth, Devon
  - Pfizer Investigational Site, Bournemouth, Dorset
  - Pfizer Investigational Site, Angus, Dundee
  - Pfizer Investigational Site, Central Milton Keyne, England
  - Pfizer Investigational Site, Lancaster, England
  - Pfizer Investigational Site, Surrey, England
  - Pfizer Investigational Site, Wishaw, Lanarkshire, England
  - Pfizer Investigational Site, Leigh-on-Sea, Essex
  - Pfizer Investigational Site, Newport, gWENT
  - Pfizer Investigational Site, Letchworth Garden City, Hertfordshire
  - Pfizer Investigational Site, Canterbury, Kent
  - Pfizer Investigational Site, Whitstable, Kent
  - Pfizer Investigational Site, Blackpool, Lancashire
  - Pfizer Investigational Site, Spalding, Lincolnshire
  - Pfizer Investigational Site, Bangor, Belfast, Northern Ireland
  - Pfizer Investigational Site, Coatbridge, Scotland
  - Pfizer Investigational Site, Glasgow, Scotland
  - Pfizer Investigational Site, Frome, Somerset
  - Pfizer Investigational Site, Stairfoot, Barnsley, South Yorkshire
  - Pfizer Investigational Site, Weybridge, Surrey
  - Pfizer Investigational Site, Leeds, West Yorkshire
  - Pfizer Investigational Site, Sheffield, Yorkshire
  - Pfizer Investigational Site, Aberdeen
  - Pfizer Investigational Site, Berkshire
  - Pfizer Investigational Site, Cambridge
  - Pfizer Investigational Site, Canterbury
  - Pfizer Investigational Site, Coventry
  - Pfizer Investigational Site, Dorking
  - Pfizer Investigational Site, Dundee
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Hertfordshire
  - Pfizer Investigational Site, Kent
  - Pfizer Investigational Site, Leeds
  - Pfizer Investigational Site, Newcastle upon Tyne
  - Pfizer Investigational Site, Nottingham
  - Pfizer Investigational Site, Rochdale
  - Pfizer Investigational Site, Shrewsbury
  - Pfizer Investigational Site, Stourbridge
  - Pfizer Investigational Site, Swanley
  - Pfizer Investigational Site, Swindon
- Pfizer Investigational Site

REFERENCES:
- [Derived] Richard Hobbs FD, Gensini G, John Mancini GB, Manolis AJ, Bauer B, Genest J, Feldman RD, Harvey P, Jenssen TG, da Silva PM; JEWEL Study Group. International open-label studies to assess the efficacy and safety of single-pill amlodipine/atorvastatin in attaining blood pressure and lipid targets recommended by country-specific guidelines: the JEWEL programme. Eur J Cardiovasc Prev Rehabil. 2009 Aug;16(4):472-80. doi: 10.1097/HJR.0b013e32832b63f5. PMID 19407658
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3841018&StudyName=Open+Label+Study+Assessing+Effectiveness+Of+Amlodipine%2FAtorvastatin+In+Subjects+With+Hypertension+and+Dyslipidaemia+